CLINICAL TRIAL: NCT06059781
Title: Combined Effects of Auditory and Visual Rhythmical Cueing on Lower Limb Sensorimotor Recovery and Gait Parameters in Patients With Hemiplegia
Brief Title: Effects of Auditory and Visual Cueing on Sensorimotor Recovery and Gait in Hemiplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Sehrish Naureen
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Hemiplegia
Keywords: auditory, visual, sensorimotor, hemiplegia, gait
MeSH Terms: conditions — Hemiplegia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhtyhmical auditory stimulation and Visual cues (Experimental group) (Experimental): For auditory stimulation, walking exercises are performed on a flat floor walking path without rhythmic or musical influence. Rhythmical auditory stimulation (RAS) is produced by using Metronome App on a mobile phone.
  For visual stimulation, white chalk will use to draw visual signals on the ground. For gait recovery, a 10-meter walkway will draw on the floor with parallel lines 2.5cm broad and 90cm long. Interline distance will maintain at 110% of the length of the initial step.
  Routine rehablitation treatment includes a range of motion exercises for the lower extremity, passive stretching of tight muscles and conventional march exercises including marching, forward, backward and sideways walking.
  Experimental group will be treated for 45 minutes per session, 3 days per week for 6 weeks.
  Interventions: Other: Rhtyhmical auditory stimulation and Visual cues (Experimental group)
- Rhtyhmical auditory stimulation (control group) (Other): For auditory stimulation, walking exercises are performed on a flat floor walking path without rhythmic or musical influence. Rhythmical auditory stimulation (RAS) is produced by using Metronome App on a mobile phone.
  Routine rehablitation treatment includes a range of motion exercises for the lower extremity, passive stretching of tight muscles and conventional march exercises including marching, forward, backward and sideways walking.
  Control group will be treated for 45 minutes per session, 3 days per week for 6 weeks.
  Interventions: Other: Rhtyhmical auditory stimulation (Control group)

INTERVENTIONS:
Other: Rhtyhmical auditory stimulation and Visual cues (Experimental group) — For auditory stimulation, walking exercises are performed on a flat floor walking path without rhythmic or musical influence. Rhythmical auditory stimulation (RAS) is produced by using Metronome App on a mobile phone.
  For visual stimulation, white chalk will use to draw visual signals on the ground. For gait recovery, a 10-meter walkway will draw on the floor with parallel lines 2.5cm broad and 90cm long. Interline distance will maintain at 110% of the length of the initial step.
  Routine recovery treatment includes a range of motion exercises for the lower extremity, passive stretching of tight muscles and conventional march exercises including marching, forward, backward and sideways walking.
  Experimental group will be treated for 45 minutes per session, 3 days per week for 6 weeks.
  Arms: Rhtyhmical auditory stimulation and Visual cues (Experimental group)
Other: Rhtyhmical auditory stimulation (Control group) — For auditory stimulation, walking exercises are performed on a flat floor walking path without rhythmic or musical influence. Rhythmical auditory stimulation (RAS) is produced by using Metronome App on a mobile phone.
  Routine recovery treatment includes a range of motion exercises for the lower extremity, passive stretching of tight muscles and conventional march exercises including marching, forward, backward and sideways walking.
  Control group will be treated for 45 minutes per session, 3 days per week for 6 weeks.
  Arms: Rhtyhmical auditory stimulation (control group)

SUMMARY:
Stroke is also known as a brain attack, happens when a blood vessel in the brain breaks or when something stops the flow of blood to a specific area of the brain. Parts of the brain undergo damage or die in either case. Stroke victims may experience permanent brain damage, long-term disability or even death. The main objective of this study is to evaluate the impact of combined auditory and visual rhythmical cueing on lower limb sensorimotor recovery and gait parameters in patients with hemiplegia. It will be a randomized controlled trial. In this study 28 patients will be recruited through non probability convenience sampling technique. The patients fulfilling inclusion and exclusion criteria will be randomly divided into experimental group (n=14) and control group (n=14) by using computer engendered in blocks by using a basic number generator. Distribution will be concealed by the sealed envelope method. Baseline treatment will be given to both groups.

Baseline treatment includes a range of motion exercises for the lower extremity, passive stretching of tight muscles and conventional march exercises including marching, forward, backward and sideways walking. Conventional training will be given for 15 minutes, 3 sessions per week for 4 weeks. Experimental group (n=14) will be treated with auditory stimulation and visual cues. All participants will undergo the training for 45 minutes per session, 3 days per week for 4 weeks. The control group (n=14) will be treated with auditory stimulation only. All participants will undergo the training for 45 minutes per session, 3 days per week for 4 weeks.

Subjective tool for sensory assessment includes Fugl-Meyer Assessment (FMA) for the lower extremity (LE) tool. For gait, it includes Dynamic Gait Index (DGI) tool. Objective tools will include cadence, gait velocity/walking speed, stride length, step length, step width, stride length symmetry ratio and step length symmetry ratio. Data will be analyzed by using SPSS (Statistical Package for Social Sciences) 23 version.

DETAILED DESCRIPTION:
A neurological condition known as a stroke is characterized by blood vessel obstruction. Brain clots prevent blood from flowing properly, obstructing arteries and causing blood vessels to burst, which causes bleeding. The abrupt death of brain cells due to a lack of oxygen occurs when the arteries leading to the brain are ruptured during a stroke . Stroke subtypes can be categorized as ischemic or hemorrhagic depending on the etiology. The majority of stroke cases (80-87%) are ischemic strokes, which can be either focal (caused by thrombosis, cardio-embolism, or atherosclerosis and platelets plugging an artery) or global (caused by a complete reduction in blood flow to the brain during a cardiac arrest). Ischemic stroke can also be lethal or not. On the other side, a blood vessel rupture results in hemorrhagic stroke . During a transient ischemic attack (TIA), arterial supply to brain tissue is temporarily cut off, resulting in focal neurologic symptoms such as hemiparesis, but spontaneous flow restoration leads to symptom relief without long-term tissue damage . Gehan M. Ahmed1, Ebtesam M. Fahmy (2023) did an RCT (randomized control trial) study in which they recruited 30 male stroke patients. Group A (control group) was treated with strengthening exercises for weak upper and lower limb, stretching exercises for lower extremity muscles, weight bearing on affected side and treadmill exercises for 6 weeks. While group B (experimental group) had rhythmical auditory stimulation (RAS) in addition with treadmill training exercise. Results of this study showed that post treatment improvement in gait parameters was significantly higher in the study group compared to the controls.

Xin Li1, Lu Wang (2022) did a controlled study in which they enrolled 24 stroke patients with severe upper limb motor deficits. One group (n=12) was treated with combined conventional training and sensorimotor rhythm-based brain computer interference (SMR-BCI) with an audio cue, motor observation with multisensory feedback for rehabilitation of upper limb. The second group(n=12) was treated with conventional treatment only. Results of this study concluded that the first group which was treated with combined conventional and (SMR-BCI) with auditory cues, motor observation with sensory feedback might promote long lasting upper limb improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 45-65 years

  * Both male and female genders
  * Clinically diagnosed of stroke referred by Neuro physician
  * Patients in the chronic stage after 6 months of stroke can walk 10 meters independently.
  * Patients with anterior cerebral artery (ACA) and middle cerebral artery (MCA) involvement with the affected side being the dominant side
  * Those with Brunnstrom's recovery stages 3 and 4 will take part
  * Patients with Mini-Mental State Examination (MMS) score greater than 16.
  * According to Modified Ashworth Scale, patients of grades 1 and 1+ will be included. Muscles that go into the spasticity include hip adductors, knee flexors and ankle plantar flexors

Exclusion Criteria:

* Patients with dementia, depression or productive psychosis will not include.

  * Patients having any visual or auditory impairment will be excluded.
  * Patients with foot drop
  * Recurrent transient ischemic attack (TIA)
  * Patients with recurrent stroke

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment FMA (LE) | Changes from baseline Fugl-Meyer Assessment FMA (LE) at 3rd week and after 6 weeks
  FMA is used to assess sensorimotor function which consists of maximum 28 points for lower extremity and 6 points for speed and coordination. The total summed score of 34 points indicates normal function. Higher the score more is the independence.
Dynamic Gait Index (DGI) | Changes from baseline Dynamic Gait Index (DGI) at 3rd week and after 6 weeks
  DGI is composed of a total of 8 items. Total score is 24. In total, a score of less than 19/24 is predictive of falls in the elderly. A score of >22 signifies a safe ambulator.
Cadence | Changes from baseline Cadence at 3rd week and after 6 weeks
  Number of steps taken per unit time
Gait velocity/Walking speed | Changes from baseline Gait velocity/Walking speed at 3rd week and after 6 weeks
  10 min walk test
Stride length | Changes from baseline Stride length at 3rd week and after 6 weeks
  Distance between successive ground contacts of the same foot by using measuring tape.
Step length | Changes from baseline Step length at 3rd week and after 6 weeks
  Distance between successive ground contact of the opposite foot by using measuring tape.
Step width | Changes from baseline Step width at 3rd week and after 6 weeks
  Transverse linear distance between two successive feet from the centers of heels by using measuring tape.
Step length symmetry ratio | Changes from baseline Step length symmetry ratio at 3rd week and after 6 weeks
  It will be calculated by dividing step length of paretic limb to non-paretic limb.
Stride length symmetry ratio | Changes from baseline Stride length symmetry ratio at 3rd week and after 6 weeks
  It will be calculated by dividing the stride length of paretic limb to non-paretic limb.

CONTACTS AND LOCATIONS:
Overall Officials: Sehrish Naureen, MSPT-NM, Principal Investigator — Riphah International University
Locations (1):
- Tehreem Mukhtar, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No